CLINICAL TRIAL: NCT04882241
Title: A Phase III, Randomized, Double-Blind, Clinical Trial of Pembrolizumab (MK-3475) Plus Chemotherapy (XP or FP) Versus Placebo Plus Chemotherapy (XP or FP) as Neoadjuvant/Adjuvant Treatment for Subjects With Gastric and Gastroesophageal Junction (GEJ) Adenocarcinoma (KEYNOTE-585)
Brief Title: Study of Pembrolizumab (MK-3475) Plus Chemotherapy Versus Placebo Plus Chemotherapy in Participants With Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma (MK-3475-585/KEYNOTE-585)-China Extension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3475-585 China Extension; MK-3475-585 (Other: MSD); 173786 (Registry Identifier: JAPIC); KEYNOTE-585 (Other: MSD); PHRR200226-002534 (Registry Identifier: PHRR Research Registration)
Record Dates: First submitted 2021-05-07; First posted 2021-05-11 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Stomach Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Saline Solution; Cisplatin; Capecitabine; Fluorouracil; Docetaxel; Oxaliplatin; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Pembrolizumab+XP/FP (Experimental): XP=cisplatin+capecitabine and FP=cisplatin+5-fluorouracil. Neoadjuvant: Prior to surgery, participants receive 3 cycles of pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets twice each day (BID) on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and 5-fluorouracil (5FU) via continuous IV infusion on Days 1 to 5 of each 3-week cycle.
  Adjuvant: 4 to 10 weeks post-surgery, participants receive pembrolizumab 200 mg via IV infusion on Day 1 Q3W PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets BID on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and 5FU via continuous IV infusion on Days 1 to 5 of each 3-week cycle for up to 3 cycles.
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: Capecitabine; Drug: 5-fluorouracil
- Placebo+XP/FP (Placebo Comparator): Neoadjuvant: Prior to surgery, participants receive 3 cycles of placebo (normal saline solution) via IV infusion on Day 1 Q3W PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets BID on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and 5FU via continuous IV infusion on Days 1 to 5 of each 3-week cycle.
  Adjuvant: 4 to 10 weeks post-surgery, participants receive placebo via IV infusion on Day 1 Q3W PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets BID on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and 5FU via continuous IV infusion on Days 1 to 5 of each 3-week cycle for up to 3 cycles.
  Interventions: Drug: Placebo; Drug: Cisplatin; Drug: Capecitabine; Drug: 5-fluorouracil
- Pembrolizumab+FLOT Cohort (Experimental): FLOT=docetaxel+oxaliplatin+5FU+leucovorin (calcium folinate). Neoadjuvant: Prior to surgery, participants receive 3 cycles of pembrolizumab 200 mg via IV infusion on Day 1 Q3W PLUS docetaxel 50 mg/m^2 via IV infusion, oxaliplatin 85 mg/m^2 via IV infusion, 5FU 2600 mg/m^2 via IV infusion, and leucovorin (calcium folinate) 200 mg/m^2 via IV infusion Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3) for 4 administrations.
  Adjuvant: 4 to 10 weeks postsurgery, participants receive pembrolizumab 200 mg via IV infusion Day 1 Q3W for up to 11 cycles PLUS docetaxel 50 mg/m^2, oxaliplatin 85 mg/m^2, 5FU 2600 mg/m^2, and leucovorin 200 mg/m^2 Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3) for 4 administrations.
  Interventions: Biological: Pembrolizumab; Drug: 5-fluorouracil; Drug: Docetaxel; Drug: Oxaliplatin; Drug: Leucovorin
- Placebo+FLOT Cohort (Placebo Comparator): Neoadjuvant: Prior to surgery, participants receive 3 cycles of placebo (normal saline solution) via IV infusion on Day 1 Q3W PLUS docetaxel 50 mg/m^2 via IV infusion, oxaliplatin 85 mg/m^2 via IV infusion, 5FU 2600 mg/m^2 via IV infusion, and leucovorin 200 mg/m^2 via IV infusion Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3) for 4 administrations.
  Adjuvant: 4 to 10 weeks postsurgery, participants receive placebo via IV infusion on Day 1 Q3W PLUS docetaxel 50 mg/m^2 via IV infusion, oxaliplatin 85 mg/m^2 via IV infusion, 5FU 2600 mg/m^2 via IV infusion, and leucovorin 200 mg/m^2 via IV infusion Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3) for 4 administrations.
  Interventions: Drug: Placebo; Drug: 5-fluorouracil; Drug: Docetaxel; Drug: Oxaliplatin; Drug: Leucovorin

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab+FLOT Cohort; Pembrolizumab+XP/FP
Drug: Placebo — IV infusion
  Other Names: Normal saline solution
  Arms: Placebo+FLOT Cohort; Placebo+XP/FP
Drug: Cisplatin — IV infusion
  Other Names: PLATINOL®
  Arms: Pembrolizumab+XP/FP; Placebo+XP/FP
Drug: Capecitabine — Oral tablets
  Other Names: XELODA®
  Arms: Pembrolizumab+XP/FP; Placebo+XP/FP
Drug: 5-fluorouracil — IV infusion
  Other Names: ADRUCIL®; 5FU
Drug: Docetaxel — IV infusion
  Other Names: TAXOTERE®
  Arms: Pembrolizumab+FLOT Cohort; Placebo+FLOT Cohort
Drug: Oxaliplatin — IV infusion
  Other Names: ELOXATIN®
  Arms: Pembrolizumab+FLOT Cohort; Placebo+FLOT Cohort
Drug: Leucovorin — IV infusion
  Other Names: WELLCOVORIN®
  Arms: Pembrolizumab+FLOT Cohort; Placebo+FLOT Cohort

SUMMARY:
The purpose of this study is to evaluate the efficacy of pembrolizumab (MK-3745) in the neoadjuvant (prior to surgery) or adjuvant (after surgery) treatment of previously untreated Chinese adults with gastric and gastroesophageal junction (GEJ) adenocarcinoma. No formal hypothesis testing will be done.

DETAILED DESCRIPTION:
The China extension study will include participants previously enrolled in China in the global study for MK-3475-585 (NCT03221426) plus those enrolled during the China extension enrollment period. A total of approximately 120 Chinese participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Has previously untreated localized gastric or gastroesophageal junction (GEJ) adenocarcinoma as defined by T3 or greater primary lesion or the presence of any positive nodes - N+ (clinical nodes) without evidence of metastatic disease.
* Plans to proceed to surgery following pre-operative chemotherapy based on standard staging studies per local practice.
* Is willing to provide tissue from a tumor lesion at baseline and at time of surgery.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1 within 3 days prior to the first dose of study treatment.
* Has adequate organ function.
* Male participants of childbearing potential must agree to use an adequate method of contraception for the course of the study through 180 days after the last dose of chemotherapy.
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 180 days after the last dose of chemotherapy or through 120 days after the last dose of pembrolizumab, whichever is greater.
* Has life expectancy of greater than 6 months.

Exclusion Criteria:

* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has received prior therapy with an anti-programmed cell death protein-1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (i.e., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], tumor necrosis factor receptor superfamily member 4 [OX-40], necrosis factor receptor superfamily member 9 [CD137]) or has previously participated in a Merck pembrolizumab (MK-3475) clinical trial.
* Has received prior systemic anti-cancer therapy including investigational agents for the current malignancy.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior the first dose of study treatment.
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ that have undergone potentially curative therapy are not excluded.
* Has a known severe hypersensitivity (≥ Grade 3) to pembrolizumab, its active substance and/or any of its excipients, or to any of the study chemotherapy agents and/or to any of their excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of Hepatitis B or known active Hepatitis C virus infection.
* Has a known history of active tuberculosis (TB).
* Female participants who are pregnant or breastfeeding or expecting to conceive children within the projected duration of the study, starting with the screening visit through180 days after the last dose of chemotherapy or through 120 days after the last dose of pembrolizumab, whichever is greater.
* Male participants who are expecting to father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of chemotherapy.
* Has had an allogenic tissue/solid organ transplant.
* Has received a live vaccine within 30 days prior to the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2025-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (20):
- China (20):
  - Afflilated Hospital of Bengbu Medical College-Surgical Oncology (Site 0638), Bengbu, Anhui
  - Beijing Friendship Hospital ( Site 0637), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 0221), Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital ( Site 0230), Fuzhou, Fujian
  - Fujian Medical University Union Hospital-1 Bingfanglou-Gastric Surgery Department (Site 0632), Fuzhou Fujian, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University (Site 0635), Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University ( Site 0224), Guangzhou, Guangdong
  - Fourth Hospital of Hebei Medical University ( Site 0633), Shijiazhuang, Hebei
  - Henan Cancer Hospital (Site 0227), Zhengzhou, Henan
  - The Affiliated Hospital of Xuzhou Medical College-Oncology ( Site 0645), Xuzhou, Jiangsu
  - The First Hospital of Jilin University-Gastrointestinal Surgery ( Site 0234), Changchun, Jilin
  - Tangdu Hospital of Fourth Military Medical University of Chinese People's Liberation Army ( Site 0647), Xi'an, Shaanxi
  - Shandong Provincial Hospital-Gastrointestinal Surgery ( Site 0640), Jinan, Shandong
  - The Affiliated Hospital of Qingdao University ( Site 0636), Qingdao, Shandong
  - Renji Hospital Shanghai Jiao Tong University School of Medicine ( Site 0642), Shanghai, Shanghai Municipality
  - Sichuan Cancer hospital, Chengdu, Sichuan
  - Zhejiang Provincial People's Hospital-Oncology (Site 0656), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0231), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital ( Site 0233), Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University (Site 0652), Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 120 participants were included in the China subpopulation. At the time of the primary analysis data cut-off, 94 participants are ongoing in the study. The FLOT cohort was not enrolled in China per specifications in the protocol Supplemental Statistical Analysis Plan (sSAP) amendment and no data were collected for the FLOT cohort in China.
Groups:
- Pembrolizumab + XP/FP: XP=cisplatin+capecitabine and FP=cisplatin+5-fluorouracil. Neoadjuvant: Prior to surgery, participants receive 3 cycles of pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets twice each day (BID) on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and 5-fluorouracil (5FU) via continuous IV infusion on Days 1 to 5 of each 3-week cycle.
  Adjuvant: 4 to 10 weeks post-surgery, participants receive pembrolizumab 200 mg via IV infusion on Day 1 Q3W PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets BID on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and 5FU via continuous IV infusion on Days 1 to 5 of each 3-week cycle for up to 3 cycles.
- Placebo + XP/FP: Neoadjuvant: Prior to surgery, participants receive 3 cycles of placebo (normal saline solution) via IV infusion on Day 1 Q3W PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets BID on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and 5FU via continuous IV infusion on Days 1 to 5 of each 3-week cycle.
  Adjuvant: 4 to 10 weeks post-surgery, participants receive placebo via IV infusion on Day 1 Q3W PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets BID on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and 5FU via continuous IV infusion on Days 1 to 5 of each 3-week cycle for up to 3 cycles.
- Pembrolizumab + FLOT Cohort: FLOT=docetaxel+oxaliplatin+5FU+leucovorin (calcium folinate). Neoadjuvant: Prior to surgery, participants receive 3 cycles of pembrolizumab 200 mg via IV infusion on Day 1 Q3W PLUS docetaxel 50 mg/m^2 via IV infusion, oxaliplatin 85 mg/m^2 via IV infusion, 5FU 2600 mg/m^2 via IV infusion, and leucovorin (calcium folinate) 200 mg/m^2 via IV infusion Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3) for 4 administrations.
  Adjuvant: 4 to 10 weeks postsurgery, participants receive pembrolizumab 200 mg via IV infusion Day 1 Q3W for up to 11 cycles PLUS docetaxel 50 mg/m^2, oxaliplatin 85 mg/m^2, 5FU 2600 mg/m^2, and leucovorin 200 mg/m^2 Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3) for 4 administrations.
- Placebo + FLOT Cohort: Neoadjuvant: Prior to surgery, participants receive 3 cycles of placebo (normal saline solution) via IV infusion on Day 1 Q3W PLUS docetaxel 50 mg/m^2 via IV infusion, oxaliplatin 85 mg/m^2 via IV infusion, 5FU 2600 mg/m^2 via IV infusion, and leucovorin 200 mg/m^2 via IV infusion Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3) for 4 administrations.
  Adjuvant: 4 to 10 weeks postsurgery, participants receive placebo via IV infusion on Day 1 Q3W PLUS docetaxel 50 mg/m^2 via IV infusion, oxaliplatin 85 mg/m^2 via IV infusion, 5FU 2600 mg/m^2 via IV infusion, and leucovorin 200 mg/m^2 via IV infusion Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3) for 4 administrations.
Period: Overall Study
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP | Pembrolizumab + FLOT Cohort | Placebo + FLOT Cohort
Started | 59 | 61 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 59 | 61 | 0 | 0
Not completed — Ongoing in study | 46 | 48 | 0 | 0
Not completed — Death | 13 | 13 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The FLOT cohort was not enrolled in China per specifications in the protocol Supplemental Statistical Analysis Plan (sSAP) amendment and no data were collected for the FLOT cohort in China.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP | Pembrolizumab + FLOT Cohort | Placebo + FLOT Cohort | Total
Number analyzed (Participants) | 59 | 61 | 0 | 0 | 120
Age, Customized [Count of Participants; unit: Participants]
  Adults (between 18 and 64 years) | 38 | 35 | 0 | 0 | 73
  From 65 to 84 years | 21 | 26 | 0 | 0 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 0 | 0 | 25
  Male | 43 | 52 | 0 | 0 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 59 | 61 | 0 | 0 | 120
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 59 | 61 | 0 | 0 | 120
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Tumor Staging [Count of Participants; unit: Participants] — Participants were categorized by tumor stage based on American Joint Committee on Cancer (AJCC) staging guidelines. The lower the cancer stage, the less the cancer has spread. Stages can range from I to IVd. 'a' describes less aggressive (slower growing) cancer, while 'd' describes more aggressive (faster growing) cancer within a numeric stage.
  Participants
    Stage II | 8 | 7 | 0 | 0 | 15
    Stage III | 49 | 48 | 0 | 0 | 97
    Stage IVa | 2 | 6 | 0 | 0 | 8
Geographic Region [Count of Participants; unit: Participants] — Participants were categorized according to geographic region of site.
  Participants
    Asia | 59 | 61 | 0 | 0 | 120

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) Per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms
Description: EFS is based on RECIST 1.1 as assessed by the investigator and is defined as the time from randomization to the first of the following events: radiographic disease progression per RECIST 1.1; local or distant recurrence as assessed by computer tomography (CT) scan or biopsy if indicated (for participants who are disease free after surgery); clinical progression as evidenced by peritoneal carcinomatosis confirmed by preoperative laparoscopy or laparotomy (for participants who are confirmed to be free of peritoneal involvement by laparoscopy at screening); or death due to any cause. A second primary malignancy, or radiographic progressive disease (PD) during the neoadjuvant phase that does not preclude successful surgery (i.e., disease free after surgery), are not considered EFS events.
Time Frame: Up to approximately 42 months
Population: The analysis population consisted of all randomized participants in the Pembrolizumab+XP/FP and Placebo+XP/FP treatment arms, as pre-specified per protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP
Number analyzed (Participants) | 59 | 61
Months | NA [15.2 to NA] — NA = Median and upper limit were not reached at time of data cut-off due to insufficient number of participants with an event | 36.5 [15.5 to NA] — NA = Upper limit was not reached at time of data cut-off due to insufficient number of participants with an event
Statistical Analysis 1: Comparison: Pembrolizumab + XP/FP vs Placebo + XP/FP; Test type: Other; p = 0.39528, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.50 to 1.70] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

2. Primary Outcome: Pathological Complete Response (pathCR) Rate - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms
Description: PathCR rate is defined as the percentage of participants having a pathCR. pathCR is defined as no invasive disease within an entirely submitted and evaluated gross lesion, and histologically negative nodes.
Time Frame: Up to approximately 9 weeks following completion of neoadjuvant treatment (up to Study Week 18)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Pembrolizumab + XP/FP: XP=cisplatin+capecitabine and FP=cisplatin+5- fluorouracil. Neoadjuvant: Prior to surgery, participants receive 3 cycles of pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets twice each day (BID) on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and 5-fluorouracil (5FU) via continuous IV infusion on Days 1 to 5 of each 3-week cycle.
  Adjuvant: 4 to 10 weeks post-surgery, participants receive pembrolizumab 200 mg via IV infusion on Day 1 Q3W PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets BID on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and 5FU via continuous IV infusion on Days 1 to 5 of each 3-week cycle for up to 3 cycles.
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP
Number analyzed (Participants) | 59 | 61
Percentage of Participants | 6.8 [1.9 to 16.5] | 4.9 [1.0 to 13.7]
Statistical Analysis 1: Comparison: Pembrolizumab + XP/FP vs Placebo + XP/FP; Test type: Other; p = 0.33244, Miettinen and Nurminen; Based on unstratified Miettinen & Nurminen method; Difference in Percentage = 1.9, 95% CI 2-sided [-7.7 to 12.0]

3. Primary Outcome: Overall Survival (OS) - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms
Description: OS is defined as the time from randomization to death due to any cause. OS is presented for the Pembrolizumab+XP/FP and Placebo+XP/FP treatment arms.
Time Frame: Up to approximately 42 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP
Number analyzed (Participants) | 59 | 61
Months | NA [NA to NA] — NA = Median, lower limit, and upper limit were not reached at time of data cut-off due to insufficient number of participants with an event | NA [25.8 to NA] — NA = Median and upper limit were not reached at time of data cut-off due to insufficient number of participants with an event
Statistical Analysis 1: Comparison: Pembrolizumab + XP/FP vs Placebo + XP/FP; Test type: Other; p = 0.52903, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.48 to 2.22] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

4. Primary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs) - Pembrolizumab+FLOT and Placebo+FLOT Cohorts
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The FLOT cohort was not enrolled in China per specifications in the protocol Supplemental Statistical Analysis Plan (sSAP) amendment and no data were collected for the FLOT cohort in China.
Time Frame: Up to approximately 42 months
Population: The FLOT cohort was not enrolled in China per specifications in the protocol sSAP amendment and no data were collected for the FLOT cohort in China.
Arm/Group | Pembrolizumab + FLOT Cohort | Placebo + FLOT Cohort
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE) - Pembrolizumab+FLOT and Placebo+FLOT Cohorts
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The FLOT cohort was not enrolled in China per specifications in the protocol sSAP amendment and no data were collected for the FLOT cohort in China.
Time Frame: Up to approximately 17 months
Population: as for outcome 4
Arm/Group | Pembrolizumab + FLOT Cohort | Placebo + FLOT Cohort
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs) - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms Separately and in Combination With the Pembrolizumab+FLOT and Placebo+FLOT Cohorts
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience at least one AE is presented for Pembrolizumab+XP/FP and Placebo+XP/FP treatment arms. The FLOT cohort was not enrolled in China per specifications in the protocol Supplemental Statistical Analysis Plan (sSAP) amendment and no data were collected for the FLOT cohort in China. There is no FLOT cohort in China to combine with XP/FP arms.
Time Frame: Up to approximately 42 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment. The FLOT cohort was not enrolled in China per specifications in the protocol sSAP amendment and no data were collected for the FLOT cohort in China. There is no FLOT cohort in China to combine with XP/FP arms.
Measure: Count of Participants; unit: Participants
Groups:
- Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined: FLOT=docetaxel+oxaliplatin+5FU+leucovorin (calcium folinate). Neoadjuvant and adjuvant pembrolizumab+XP/FP and neoadjuvant and adjuvant pembrolizumab+FLOT Cohort treatment arms combined
- Placebo + XP/FP and Placebo + FLOT Cohort Combined: Neoadjuvant and adjuvant placebo+XP/FP and neoadjuvant and adjuvant placebo+FLOT Cohort treatment arms combined
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP | Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined | Placebo + XP/FP and Placebo + FLOT Cohort Combined
Number analyzed (Participants) | 59 | 61 | 0 | 0
Participants | 59 | 61 |  |

7. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE) - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms Separately and in Combination With the Pembrolizumab+FLOT and Placebo+FLOT Cohorts
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be presented for Pembrolizumab+XP/FP and Placebo+XP/FP treatment arms. The FLOT cohort was not enrolled in China per specifications in the protocol sSAP amendment and no data were collected for the FLOT cohort in China. There is no FLOT cohort in China to combine with XP/FP arms.
Time Frame: Up to approximately 23 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP | Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined | Placebo + XP/FP and Placebo + FLOT Cohort Combined
Number analyzed (Participants) | 59 | 61 | 0 | 0
Participants | 12 | 8 |  |

8. Secondary Outcome: Disease-free Survival (DFS) Per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms
Description: DFS is defined as the time from post-surgery baseline scan until the first occurrence of local/distant recurrence or death from any cause and is based on RECIST 1.1 as assessed by the investigator.
Time Frame: Up to approximately 42 months
Population: The analysis population consisted of all randomized participants in the Pembrolizumab+XP/FP and Placebo+XP/FP treatment arms who had surgery, as pre-specified per protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP
Number analyzed (Participants) | 42 | 42
Months | NA [15.2 to NA] — NA = Median and upper limit were not reached at time of data cut-off due to insufficient number of participants with an event | 33.1 [16.6 to NA] — NA = Upper limit was not reached at time of data cut-off due to insufficient number of participants with an event
Statistical Analysis 1: Comparison: Pembrolizumab + XP/FP vs Placebo + XP/FP; Test type: Other; p = 0.34632, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.34 to 2.05] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

9. Secondary Outcome: Overall Survival (OS) - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms in Combination With the Pembrolizumab+FLOT and Placebo+FLOT Cohorts
Description: OS is defined as the time from randomization to death due to any cause. The FLOT cohort was not enrolled in China per specifications in the protocol sSAP amendment and no data were collected for the FLOT cohort in China. There is no FLOT cohort in China to combine with XP/FP arms.
Time Frame: Up to approximately 42 months
Population: The FLOT cohort was not enrolled in China per specifications in the protocol sSAP amendment and no data were collected for the FLOT cohort in China. There is no FLOT cohort in China to combine with XP/FP arms.
Groups:
- Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined: Neoadjuvant and adjuvant pembrolizumab+XP/FP and neoadjuvant and adjuvant pembrolizumab+FLOT Cohort treatment arms combined
Arm/Group | Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined | Placebo + XP/FP and Placebo + FLOT Cohort Combined
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Event-free Survival (EFS) Per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms in Combination With the Pembrolizumab+FLOT and Placebo+FLOT Cohorts
Description: EFS is based on RECIST 1.1 as assessed by the investigator and is defined as the time from randomization to the first of the following events: radiographic disease progression per RECIST 1.1; local or distant recurrence as assessed by CT scan or biopsy if indicated (for participants who are disease free after surgery); clinical progression as evidenced by peritoneal carcinomatosis confirmed by preoperative laparoscopy or laparotomy (for participants who are confirmed to be free of peritoneal involvement by laparoscopy at screening); or death due to any cause. A second primary malignancy, or radiographic progressive disease (PD) during the neoadjuvant phase that does not preclude successful surgery (i.e., disease free after surgery), are not considered EFS events. The FLOT cohort was not enrolled in China per specifications in the protocol sSAP amendment and no data were collected for the FLOT cohort in China. There is no FLOT cohort in China to combine with XP/FP arms.
Time Frame: Up to approximately 42 months
Population: as for outcome 9
Arm/Group | Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined | Placebo + XP/FP and Placebo + FLOT Cohort Combined
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 42 months
Description: All-Cause Mortality includes all randomized participants. Serious and Other AEs includes all randomized participants who received ≥1 dose of study treatment. The FLOT cohort was not enrolled in China per specifications in the protocol sSAP amendment and no data were collected for the FLOT cohort in China. MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs.
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP
All-Cause Mortality (participants affected / at risk) | 13/59 | 13/61
Serious Adverse Events (participants affected / at risk) | 32/59 | 30/61
Other Adverse Events (participants affected / at risk) | 59/59 | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + XP/FP (N=59) | Placebo + XP/FP (N=61)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Volvulus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 8 (9)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Ulcer (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 3 (3)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Haematological infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 3 (4)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (5) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 3 (4)
Weight decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 6 (7) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 3 (3) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + XP/FP (N=59) | Placebo + XP/FP (N=61)
Anaemia (Blood and lymphatic system disorders) | 45 (85) | 47 (85)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 6 (9) | 4 (9)
Neutropenia (Blood and lymphatic system disorders) | 4 (8) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (6) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 2 (2)
Hypothyroidism (Endocrine disorders) | 11 (17) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 6 (7) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 8 (10) | 10 (11)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 5 (5)
Constipation (Gastrointestinal disorders) | 15 (18) | 18 (18)
Diarrhoea (Gastrointestinal disorders) | 19 (24) | 7 (10)
Dyspepsia (Gastrointestinal disorders) | 6 (8) | 5 (7)
Nausea (Gastrointestinal disorders) | 45 (100) | 49 (120)
Vomiting (Gastrointestinal disorders) | 37 (72) | 31 (67)
Asthenia (General disorders) | 1 (1) | 5 (6)
Fatigue (General disorders) | 10 (11) | 5 (7)
Malaise (General disorders) | 4 (4) | 3 (4)
Pyrexia (General disorders) | 15 (18) | 10 (15)
COVID-19 (Infections and infestations) | 14 (15) | 9 (11)
Pneumonia (Infections and infestations) | 3 (3) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 8 (14) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 12 (12) | 13 (13)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Alanine aminotransferase increased (Investigations) | 17 (26) | 12 (16)
Aspartate aminotransferase increased (Investigations) | 17 (27) | 13 (15)
Blood alkaline phosphatase increased (Investigations) | 6 (6) | 0 (0)
Blood bilirubin increased (Investigations) | 6 (7) | 3 (4)
Blood creatinine increased (Investigations) | 9 (13) | 4 (4)
Blood urea increased (Investigations) | 2 (4) | 4 (8)
C-reactive protein increased (Investigations) | 4 (4) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 5 (6) | 0 (0)
Lymphocyte count decreased (Investigations) | 17 (32) | 9 (19)
Neutrophil count decreased (Investigations) | 47 (125) | 50 (171)
Platelet count decreased (Investigations) | 31 (79) | 35 (76)
SARS-CoV-2 test positive (Investigations) | 4 (4) | 4 (4)
Weight decreased (Investigations) | 23 (24) | 34 (36)
White blood cell count decreased (Investigations) | 45 (138) | 46 (168)
Decreased appetite (Metabolism and nutrition disorders) | 25 (31) | 29 (39)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (10) | 6 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (8) | 3 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 (10) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (9) | 4 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 28 (48) | 18 (24)
Hypocalcaemia (Metabolism and nutrition disorders) | 13 (19) | 9 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (35) | 13 (23)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (12) | 4 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 14 (30) | 9 (13)
Hypophosphataemia (Metabolism and nutrition disorders) | 7 (10) | 2 (4)
Hypoproteinaemia (Metabolism and nutrition disorders) | 10 (17) | 11 (16)
Malnutrition (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 7 (10) | 5 (8)
Headache (Nervous system disorders) | 3 (7) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 11 (12) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT04882241/Prot_SAP_001.pdf